CLINICAL TRIAL: NCT04544917
Title: Development of an eHealth-based Cognitive Behavioral Stress and Self-Management Intervention to Reduce Symptom Burden in HIV+ Gay and Bisexual Men Who Have Sex With Men (MSM) Treated for Non-Metastatic Cancer
Brief Title: SmartManage Stress Management for HIV+ Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190762
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Hiv; Stress
Keywords: Symptom burden; Cognitive behavioral stress management; Intervention development
MeSH Terms: conditions — Neoplasms; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartManage Group (Experimental): Participants in this group will receive ten 90-minute weekly therapist delivered SmartManage group sessions via video conference. Participants will have access to the SmartManage web platform, which will also guide the live intervention sessions.
  Interventions: Behavioral: SmartManage for HIV+ cancer survivors
- Educational Control Group (Active Comparator): Participants in this group will view ten weekly control content video recorded sessions.
  Interventions: Behavioral: Educational Control

INTERVENTIONS:
Behavioral: SmartManage for HIV+ cancer survivors — Ten weekly therapist delivered group sessions delivered via web conference. Sessions focus on cognitive behavioral stress management, psychoeducation, and management strategies for dual diagnosis of HIV and cancer. Participants will have access to the SmartManage web platform which has all intervention material, resources, and exercises.
  Arms: SmartManage Group
Behavioral: Educational Control — Participants in the control condition will view ten videos over ten weeks, consisting of informational and educational material relevant to cancer and HIV.
  Arms: Educational Control Group

SUMMARY:
The purpose of this study is to design and refine a web-based platform developed for managing symptom burden in men who have sex who are HIV+ cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Fluent in English
3. Have evidence of at least one form of non-metastatic solid tumor cancer or blood cancer
4. Be at least 30 days post active primary cancer treatment
5. Self identify as a sexual minority cisgender man
6. Self-report having been diagnosed with HIV
7. Have reliable access to a computer/device with internet accessibility

Exclusion Criteria:

1. Have had one of the following exclusionary cancer types: Non-melanoma skin cancer, brain cancer, eye cancer, history of some form of pediatric cancer (if that is participant's only cancer diagnosis)
2. History of advanced (metastatic) cancer of any type
3. Inpatient treatment for severe mental illness in the past 12 months and/or suicidality of moderate or greater risk
4. Appears actively intoxicated or otherwise unable to provide full informed consent
5. Have any other medical condition resulting in predicted live expectancy of less than 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male sex assigned at birth and self-identify as male.
Enrollment: 32 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible SMM that agree to participate | Up to one year
  Feasibility of the intervention will be reported as the proportion of eligible sexual minority men (SMM) who agree to participate versus decline

SECONDARY OUTCOMES:
USE Questionnaire Scores | Week 10
  Acceptability of the intervention will be reported as Usefulness, Satisfaction and Ease of Use (USE) Questionnaire Scores. USE is a 30-item questionnaire with a total score ranging from 30-240 with the higher score indicating greater acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Penedo, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No